CLINICAL TRIAL: NCT03009942
Title: Nitric Oxide and Arginase Levels in Peri-Implant Tissues After Delayed Loading
Brief Title: Biochemical Mediators After Implant Loading
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Nurdan Ozmeric, Professor, Gazi University
Other Study IDs: 03/2008-19
Record Dates: First submitted 2017-01-02; First posted 2017-01-04 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Implant Loading
Keywords: nitric oxide; arginase; loading

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
This study evaluates the nitric oxide and arginase levels in patients with dental implants. Peri-implant sulcular fluid and saliva samples were collected after loading of the implants

DETAILED DESCRIPTION:
Nitric oxide (NO) metabolism is associated with the clinical inflammatory state of peri-implant tissues and also affected by the mechanic stimulus. Therefore, The NO content of PISF reflects two different measures and can serve as an indicator of peri-implant soft tissue inflammation and/or bone response to force application and loading Arginase may reduce NO production by depleting the common substrate. Thus, increased salivary arginase activities detected in periodontitis patients may cause decreased NO synthesis and lead to a decrease in the antibacterial property of saliva.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ≥ 20 teeth, no systemic diseases that could affect bone metabolism, no smoking habits, and had one or more implants

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Twenty patients with one or more implants restored with fixed crown prostheses
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-01; Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Biochemical parameters (nitric oxide and arginase) in periimplant sulcular fluid and saliva | Baseline and 1, 3 and 6 months after implant loading
  The changes in nitric oxide and arginase levels after implant loading were determined.

SECONDARY OUTCOMES:
Plaque index | Baseline and 1, 3 and 6 months after implant loading
  The changes in plaque index after implant loading. Plaque index was recorded for determining and classifying oral hygiene status.
Gingival index | Baseline and 1, 3 and 6 months after implant loading
  The changes in gingival index after implant loading. Gingival index was recorded for classifying and evaluating gingival inflammation.
Probing depth | Baseline and 1, 3 and 6 months after implant loading
  The changes in probing pocket depth after implant loading.Probing pocket depth was measured for determining periimplant health.
Bleeding on probing | Baseline and 1, 3 and 6 months after implant loading
  The changes in bleeding on probing after implant loading. Bleeding on probing was recorded for evaluating gingival inflammation.